CLINICAL TRIAL: NCT04179812
Title: Multimodal Modeling of the Knee Joint
Acronym: KneeMod
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: KneeMod ( 29BRC18.0235)
Record Dates: First submitted 2019-06-21; First posted 2019-11-27 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trial will contribute to the development of an innovative algorithm that aims to simplify and improve preoperative knee surgical decision. This will be made by automatically extracting anatomical informations from different images acquired on the patient (scanner, MRI, radiography).

DETAILED DESCRIPTION:
The source population will consist of at least 50 patients whose following modalities of images of the leg are present in the database: scanner, MRI, radiography. No restrictions on age or gender are required.

A dedicated algorithm adapting statistical models of appearance to the specific morphology of the patient acquired through an MRI and / or scanner and radios will then be developed.

ELIGIBILITY:
Inclusion Criteria:

* Patients having the 3 modality of images : scanner, MRI, radiography
* Patients having osteoarthritis or knee trauma
* Images showing the articualtion of the knee
* having formulated his non opposition

Exclusion Criteria:

* Presentation of a partial view of the knee or any view that does not allow a good segmentation of the total knee joint.
* Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Targeted patients will be those whose leg image modalities are present in the Brest University Hospital database
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2019-03-16 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Obtaining a similar knee segmentation for all patient regardless of the input image (MRI, CT or radiography) | Inclusion - Day 0
  Creation of an algorithm that will automatically segment and provide the same knee anatomical informations for all patients studied regardless of the input image.
  This multimodal modeling will be carried out via the exploitation of an active model of appearance type algorithm.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France